CLINICAL TRIAL: NCT01738191
Title: Atomoxetine Treatment for Cognitive Impairment in Parkinson's Disease (ATM-Cog)
Acronym: ATM-Cog
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Vanessa Hinson, Director, Movement Disorders Program, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATM-Cog
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Parkinson's Disease; Cognitive Impairment
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomoxetine (Active Comparator): The study drug target dose is Atomoxetine (ATM) 80 milligram (mg) per day; given as a once daily dose of an 80mg capsule. Patients will titrate up to target dose by starting on ATM 40mg capsules: 1 capsule daily for 14 days. Following study visit 3 (after 2 weeks on the titration dose), patients will increase the dose of ATM to 80mg daily.
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Patients in the placebo arm will follow the same titration schedule as those in the active arm. Patients will titrate up to target dose by starting 40mg capsules: 1 capsule daily for 14 days. Following study visit 3 (after 2 weeks on the titration dose), patients will increase the dose to 80mg daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — The study drug target dose is ATM 80mg per day; given as a once daily dose of an 80mg capsule. Patients will titrate up to target dose by starting on ATM 40mg capsules: 1 capsule daily for 14 days. Following study visit 3 (after 2 weeks on the titration dose), patients will increase the dose of ATM to 80mg daily.
  Other Names: Strattera
  Arms: Atomoxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a drug called atomoxetine for the treatment of cognitive impairment for Parkinson 's disease. Atomoxetine (ATM) is an approved drug currently on the market for the treatment of attention deficit. It works to increase the amount of norepinephrine (a chemical in the brain that helps keep us awake and alert) in our brain. ATM has not been approved by the Food and Drug Administration (FDA) to be used in the treatment of PD.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of idiopathic PD according to the United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) criteria
* Male or female subjects aged between 35 and 75 years, inclusive at the time of consent
* Hoehn & Yahr Stage I-IV
* Diagnosis of PD mild cognitive impairment (MCI), Montreal Cognitive Assessment (MoCa) score 21-25
* Stable concomitant medications for 60 days

Exclusion Criteria:

* Secondary parkinsonism or atypical parkinsonism, Prior Deep Brain Stimulation (DBS) or other brain surgery
* PD Dementia; MoCA score <21
* Presence of Psychosis, pregnancy, suicidal ideation on the Columbia Suicide Severity Rating Scale (C-SSRS) type 4 or 5 in past 3 months.
* Current treatment with anticholinergics, monoamine oxidase (MAO) inhibitors or neuroleptics (including quetiapine)
* Serious cardiac abnormalities, Narrow angle glaucoma, Pheochromocytoma, Bipolar Disorder
* Liver Function Tests (LFTs) >1.5 X upper limit of normal value

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa K Hinson, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients in the placebo arm will follow the same titration schedule as those in the active arm. Patients will titrate up to target dose by starting 40mg capsules: 1 capsule daily for 14 days. Following study visit 3 (after 2 weeks on the titration dose), patients will increase the dose to 80mg daily.
  Placebo
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 15 | 15
Completed | 11 | 14
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (6.5) | 66.7 (7.7) | 66.8 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: The Global Statistical Test Combined Information on Change From Baseline on a Battery of Standardized Executive Function Tests
Description: Patients were ranked on each outcome and ranks were summed. The mean summed-ranks were compared by treatment group by a global statistical test (GST). Higher scores indicate better performance. The total summed-ranks range from 7 - 210 (7 outcomes x N=30).
Time Frame: change from baseline and 10 weeks
Population: Intent-to-treat sample of all patients randomized.
Measure: Mean (95% Confidence Interval); unit: summed-ranks
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 15 | 15
summed-ranks | 99.5 [73.1 to 126.0] | 117.5 [98.5 to 136.4]
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; The primary comparison between ATM and placebo used O'Brien's Global Statistical Test (GST) to analyze change from baseline to 10 weeks for the set of neuropsychological measures included in the primary efficacy outcome; Test type: Superiority; p = 0.25, Global Statistical Test — two sided; df=28

2. Secondary Outcome: Change in PASAT
Description: Paced Auditory Serial Addition Test 3-second interstimulus interval | Z-score| age & education normed| range -5 to +5 Higher scores mean a better outcome.
Time Frame: change from baseline and 10 weeks
Population: Intent-to-treat sample of all patients randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | -0.96 (1.96) | 0.42 (1.22)

3. Secondary Outcome: Change in NAB: Part A
Description: Neuropsychological Assessment Battery Numbers & Letters A Efficiency | T-score| age & education normed| range 19-70
  Higher scores mean a better outcome.
Time Frame: change from baseline and 10 weeks
Population: Intent-to-treat sample of all patients randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | -0.71 (1.05) | -0.23 (1.07)

4. Secondary Outcome: Change in NAB: Part D
Description: Neuropsychological Assessment Battery Numbers & Letters D Efficiency | T-score| age & education normed| range 19-70
  Higher scores mean a better outcome.
Time Frame: change from baseline and 10 weeks
Population: Intent-to-treat sample of all patients randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | -0.35 (1.31) | -0.11 (0.75)

5. Secondary Outcome: Change in D-KEFS: Inhibition Time
Description: Delis-Kaplan Executive Function System Color-Word Inhibition Time | Scaled | age normed| range 1-16 Higher scores mean a better outcome.
Time Frame: change from baseline and 10 weeks
Population: Intent-to-treat sample of all patients randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | -0.77 (1.4) | -0.3 (1.17)

6. Secondary Outcome: Change in D-KEFS: Inhibition-Switching Time
Description: Delis-Kaplan Executive Function System Color-Word Inhibition/Switching | Scaled | age normed| range 1-16 Higher scores mean a better outcome.
Time Frame: change from baseline and 10 weeks
Population: Intent-to-treat sample of all patients randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | -0.87 (1.63) | -0.2 (1.63)

7. Secondary Outcome: Change in D-KEFS: Number-Letter Switching Time
Description: Delis-Kaplan Executive Function System Trail Making Number/Letter Switching | Scaled | age normed| range 1-16 Higher scores mean a better outcome.
Time Frame: change from baseline and 10 weeks
Population: Intent-to-treat sample of all patients randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | -0.9 (1.33) | -0.67 (1.43)

8. Secondary Outcome: Change in WAIS-IV: Digit Span
Description: Wechsler Adult Intelligence Scale, fourth edition Digit Span | Scaled | age| 1-16
  Higher scores mean a better outcome.
Time Frame: change from baseline and 10 weeks
Population: Intent-to-treat sample of all patients randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | -0.17 (0.8) | 0 (0.67)

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=15) | Placebo (N=15)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Jitters (Nervous system disorders) | 3 (3) | 1 (3)
Syncopal Episode (Cardiac disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Decreased memory (Nervous system disorders) | 0 (0) | 1 (3)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes